CLINICAL TRIAL: NCT02004847
Title: Monocenter, Randomized, Double Blinded, Intraindividual, Exploratory Study of Effectiveness and Safety of 3 Months Treatment With 2 Peak Intensities of 453nm Blue Light for the Treatment of Mild Plaque Type Psoriasis Vulgaris
Brief Title: Blue Light for Treating Psoriasis Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Electronics Nederland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PsoriasisCT02
Record Dates: First submitted 2013-11-19; First posted 2013-12-09 (Estimated); Results first posted 2015-11-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-11

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Intensity (HI) vs control (Experimental): PSO-CT02 device: Light wavelength 453nm, high intensity, compared to contralateral untreated control plaque on the same patient.
  Interventions: Device: PSO-CT02
- Low Intensity (LI) vs control (Experimental): PSO-CT02 device: Light wavelength 453nm, low intensity, compared to contralateral untreated control plaque on the same patient.
  Interventions: Device: PSO-CT02

INTERVENTIONS:
Device: PSO-CT02 — The PSO-CT02 device is a non CE marked investigational medical device that is worn on the affected skin area where it irradiates the Psoriasis plaque for 30 minutes with blue light.

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a blue light device for treating Psoriasis vulgaris. The study will compare a blue light treated plaque with an untreated control plaque. Additionally, two intensities of blue light are compared.

DETAILED DESCRIPTION:
Blue light has been shown to release bioactive nitric oxide (NO) from nitrite and nitrosated proteins found in high concentrations in the skin. This bioactive NO has many physiological functions regulating immune responses, proliferation / differentiation as well as local blood Perfusion of the skin. The study will test the PSO-CT02 device, an new investigational medical device emitting blue light with a peak wavelength of 453nm on treating localised mild Psoriasis vulgaris. It can be worn on the Skin above the effected skin area. In this study Treatment (target) and control area as well as intensity of blue light are randomized. The control area will serve as reference. 50 Patients will treat the target area daily (at least 5 times/week) at home for an initial treatment period of 4 weeks. During those 4 weeks, patients will return to the study site for safety and effectiveness assessments twice. After this initiation period patients will treat their plaque for further 8 weeks (3 times/week). This is followed by a 4 week follow up phase without treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent prior to any study mandated procedure
2. Good health according to physical examination as determined by the Investigator
3. Willing and able to comply with study requirements
4. Skin type I-IV according to Fitzpatrick
5. Mild plaque-type psoriasis vulgaris with a Psoriasis area severity index (PASI) ≤10 and Body surface area (BSA)

   ≤10 and Dermatology Life quality index (DLQI) ≤ 10 at screening.
6. Presence of two comparable psoriatic plaques suitable to be defined as study areas as follows:

   1. located on extremities (plaques located on the palms or sole of the feet are not suitable)
   2. Both areas located either on lower or upper extremity
   3. Can be located on the same extremity
   4. Distance between the two study areas > 10cm (border to border)
   5. If lesion is too large to be fully covered, partial treatment possible
7. Aged ≥ 18 years up to <75 years
8. Reliable method of contraception for women of childbearing potential (i.e. low failure rate less than 1% per year; e.g. oral contraceptives, intra-uterine device [IUD] or transdermal contraceptive patch)
9. Willing to abstain from excessive sun / UV exposure (e.g. sunbathe, solarium) during the course of the study.

Exclusion Criteria:

General

1. Inmates of psychiatric wards, prisons, or other state institutions
2. Investigator or any other team member involved directly or indirectly in the conduct of the clinical study
3. Participation in another clinical trial within the last 30 days
4. Pregnant or lactating women Medical History
5. Photodermatosis and/or Photosensitivity
6. Porphyria and/or hypersensitivity to porphyrins
7. Patients with current diagnosis of erythrodermic, exfoliative or pustular psoriasis
8. Congenital or acquired immunodeficiency
9. Patients with any of the following conditions present on the study areas: Malignoma of the skin or severe actinic damage of the skin, atypical naevi or signs of hyperpigmentation, viral (e.g. herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections and atrophic Skin
10. Patients with genetic deficiencies attached with increased sensitivity to light or increased risk to dermatologic cancer (i.e. Xeroderma pigmentosum, Cockayne Syndrome, Bloom- Syndrome)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Verena von Felbert, PD, Dr., Principal Investigator — Clinic for Dermatology and Allergology, Medical Faculty of the RWTH Aachen, Germany
Locations (1):
- Department of Dermatology and Allergology, Medical faculty of the RWTH Aachen, Aachen, Germany

REFERENCES:
- [Derived] Pfaff S, Liebmann J, Born M, Merk HF, von Felbert V. Prospective Randomized Long-Term Study on the Efficacy and Safety of UV-Free Blue Light for Treating Mild Psoriasis Vulgaris. Dermatology. 2015;231(1):24-34. doi: 10.1159/000430495. Epub 2015 Jun 2. PMID 26044167

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patient visits were conducted at the Department of Dermatology and Allergology, RWTH Aachen University Hospital. One hundred and twenty-nine patients were prescreened, 49 patients were screened and 47 enrolled in the study at the time of screening from October 2013 to June 2014.
Pre-assignment Details: Two patients were screening failures, so 47 actually started the study.
Groups:
- High Intensity (HI) vs. Control: PSO-CT02 device: Light wavelength 453nm, high intensity versus contralateral untreated control plaque on the same patient.
- Low Intensity (LI) vs. Control: PSO-CT02 device: Light wavelength 453nm, low intensity versus contralateral untreated control plaque on the same patient.
Period: Overall Study
Arm/Group | High Intensity (HI) vs. Control | Low Intensity (LI) vs. Control
Started | 24 | 23
Completed | 23 | 22
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Aanalysis Set (FAS)
Groups:
- Total: Total of all reporting groups
Arm/Group | High Intensity (HI) vs Control | Low Intensity (LI) vs Control | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 45
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.54 (13.80) | 49.09 (10.68) | 47.79 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  Germany | 24 | 23 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Visit 2) of the Local Psoriasis Area Severity Index (PASI) of the Target Area (High Intensity (HI) Group) as Compared to the Control Area at End of Treatment (Visit 7, Week 12).
Description: In this study only the "local" PASI (also called local psoriasis severity index - LPSI) was evaluated. The investigator evaluated and graded the severity of erythema, induration, and scaliness as the key symptoms of psoriasis on the study areas using the following scale:
  0 = no sign, 1 = slight, 2 = moderate, 3 = marked,4 = very marked
  A total severity score was calculated as the sum of the three symptom ratings (range 0-12 whereas 0 (best) - 12 (worst)).
Time Frame: baseline and week 12
Population: Full Analysis set (FAS)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- High Intensity (HI): PSO-CT02 device: Light wavelength 453nm, high intensity
- Control (HI): Contralateral untreated control plaque on the same patient.
Arm/Group | High Intensity (HI) | Control (HI)
Number analyzed (Participants) | 24 | 24
units on a scale | -2.38 (1.53) | -1.46 (1.59)
Statistical Analysis 1: Comparison: High Intensity (HI) vs Control (HI); Statistically analysed were the difference in change from baseline to the end of treatment (week 12) of the target plaque compared to the control plaque; Test type: Superiority or Other; p = 0.0005, t-test, 2 sided

2. Secondary Outcome: Change From Baseline of the Local Psoriasis Area Severity Index (PASI) of the Target Area (High Intensity) as Compared to the Control Area at End of Treatment During the Attack Period (Week 4, Visit 5)
Description: as for outcome 1
Time Frame: baseline and week 4
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Intensity (HI) | Control (HI)
Number analyzed (Participants) | 24 | 24
units on a scale | -1.92 (1.21) | -1.33 (1.66)
Statistical Analysis 1: Comparison: High Intensity (HI) vs Control (HI); Statistically analysed were the difference in change from baseline to the end of treatment during the attack period (week 4) of the target plaque compared to the control plaque; Test type: Superiority or Other; p = 0.0036, t-test, 2 sided

3. Secondary Outcome: Change From Week 12 of the Local Psoriasis Area Severity Index (PASI) of the Target Area (High Intensity) as Compared to the Control Area at End of Follow-up
Description: as for outcome 1
Time Frame: Week 12 and week 16
Population: Full Analysis Set (FAS); due to one drop out this number is 23 at week 12 and 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Intensity (HI) | Control (HI)
Number analyzed (Participants) | 23 | 23
units on a scale | -0.22 (1.313) | -0.43 (1.590)
Statistical Analysis 1: Comparison: High Intensity (HI) vs Control (HI); Statistically analysed were the difference in change from end of treatment (week 12, visit 7) to end of follow up (week 16, visit 8) of the target plaque compared to the control plaque; Test type: Superiority or Other; p = 0.3075, t-test, 2 sided

4. Secondary Outcome: Change From Baseline (Visit 2) of the Local Psoriasis Area Severity Index (PASI) of the Target Area (Low Intensity (LI) Group) as Compared to the Control Area by Week.
Description: as for outcome 1
Time Frame: baseline and week 4, 12, 16
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Low Intensity: PSO-CT02 device: Light wavelength 453nm, low intensity
- Control (LI): Contralateral untreated control plaque on the same patient.
Arm/Group | Low Intensity | Control (LI)
Number analyzed (Participants) | 23 | 23
units on a scale
  week 4 | -1.83 (1.557) | -0.87 (1.604)
  week 12 | -2.78 (1.347) | -2.04 (1.461)
  week 16 | -3.00 (1.447) | -2.50 (1.655)
Statistical Analysis 1: Comparison: Low Intensity vs Control (LI); Statistically analysed were the difference in change from baseline to week 4 of the target plaque compared to the control plaque; Test type: Superiority or Other; p = 0.0140, t-test, 2 sided
Statistical Analysis 2: Comparison: Low Intensity vs Control (LI); Statistically analysed were the difference in change from baseline to week 12 of the target plaque compared to the control plaque; Test type: Superiority or Other; p = 0.0064, t-test, 2 sided
Statistical Analysis 3: Comparison: Low Intensity vs Control (LI); Statistically analysed were the difference in change from baseline to week 16 of the target plaque compared to the control plaque; Test type: Superiority or Other; p = 0.1020, t-test, 2 sided

5. Secondary Outcome: Difference in Change From Baseline of Local Psoriasis Area Severity Index (PASI) Between Target and Control Area of the High Intensity (HI) Group as Compared to the Low Intensity (LI) Group
Description: In this study only the "local" PASI (also called local psoriasis severity index - LPSI) was evaluated. The investigator evaluated and graded the severity of erythema, induration, and scaliness as the key symptoms of psoriasis on the study areas using the following scale:
  0. = no sign
  1. = slight
  2. = moderate
  3. = marked
  4. = very marked A total severity score was calculated as the sum of the three symptom ratings (range 0-12).
Time Frame: baseline and week 4, 8, 16
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Low Intensity (LI): PSO-CT02 device: Light wavelength 453nm, low intensity
Arm/Group | High Intensity (HI) | Control (HI) | Low Intensity (LI) | Control (LI)
Number analyzed (Participants) | 24 | 24 | 23 | 23
units on a scale
  week 4 n=24 (HI) n=23 (LI) | -1.92 (1.213) | -1.33 (1.659) | -1.83 (1.557) | -0.87 (1.604)
  week 8 n=24 (HI) n=23 (LI) | -2.25 (1.359) | -1.50 (1.719) | -1.78 (1.650) | -1.30 (1.460)
  week 16 n=23 (HI) n=22 (LI) | -2.57 (1.619) | -1.87 (1.842) | -3.00 (1.447) | -2.50 (1.655)

6. Secondary Outcome: Change From Baseline of Erythema Evaluated by Mexameter of the Target Area of High Intensity (HI) and Low Intensity (LI) as Compared to the Control Area
Description: Erythema was measured directly after treatment. Mexameter readings ranged from 0 to 100. Higher values describe higher erythema levels.
Time Frame: baseline and week 4, 12
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- High Intensity (HI): PSO-CT02 device: Light wavelength 453nm, high intensity versus contralateral untreated control plaque on the same patient.
- Low Intensity (LI): PSO-CT02 device: Light wavelength 453nm, low intensity versus contralateral untreated control plaque on the same patient.
Arm/Group | High Intensity (HI) | Control (HI) | Low Intensity (LI) | Control (LI)
Number analyzed (Participants) | 24 | 24 | 23 | 23
arbitrary units
  4 weeks | 3.38 (13.87) | 1.00 (13.45) | 0.13 (11.90) | 2.87 (12.00)
  12 weeks | -0.38 (11.02) | -0.58 (11.82) | 5.50 (16.66) | 1.05 (9.77)

7. Secondary Outcome: Change From Week 12 (End of Treatment) of Erythema Evaluated by Mexameter of the Target Area of High Intensity (HI) and Low Intensity (LI) as Compared to the Control Area at End of Follow-up
Description: as for outcome 6
Time Frame: week 12 and week 16
Population: Full Analysis Set (FAS); due to one drop out in each group this number is 23 for HI Group and 22 for LI group at week 12 and 16
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | High Intensity (HI) | Control (HI) | Low Intensity (LI) | Control (LI)
Number analyzed (Participants) | 23 | 23 | 22 | 22
arbitrary units | -2.26 (14.08) | 2.00 (14.97) | -1.64 (12.07) | 3.23 (9.97)

8. Secondary Outcome: System Usability Scale
Description: At the end of treatment (visit 7), the usability of the investigational device was evaluated by a questionnaire presented to the patient in German. The usability was evaluated by using the System Usability Scale (SUS) which is an effective tool for assessing the usability of a device. It provides an easy-to-understand score from 0 (negative) to 100 (positive).
Time Frame: week 12
Population: Full Analysis Set (FAS); due to one drop out this number is 23 at week 12 for HI group. Only 17 of 22 patients completed the questionaire in the LI group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Intensity (HI) | Low Intensity (LI)
Number analyzed (Participants) | 23 | 17
units on a scale | 88.37 (11.62) | 88.53 (9.02)

9. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI)
Description: It is a simple 10-question validated questionnaire. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. As the change from baseline is calculated negative values in the Outcome Measure Data indicate an improvement in quality of life.
Time Frame: baseline and week 12
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Intensity (HI) | Low Intensity (LI)
Number analyzed (Participants) | 24 | 22
units on a scale | -0.75 (2.98) | -0.36 (4.18)

10. Secondary Outcome: Time to First Use of Topical Co-treatment With Vitamin D of High Intensity (HI) and Low Intensity (LI)
Time Frame: patients will be followed for the complete duration of the clinical study for 16 weeks
Population: Full Analysis Set (FAS); Not all patients requested co-use of vitamin D. Only 17 in HI group and 16 in LI group requested co-use of vitamin D
Measure: Mean (Standard Deviation); unit: days
Arm/Group | High Intensity (HI) | Low Intensity (LI)
Number analyzed (Participants) | 17 | 16
days | 46.35 (17.68) | 48.25 (26.36)

11. Secondary Outcome: Total Duration of Topical Co-treatment With Vitamin D of High Intensity (HI) and Low Intensity (LI)
Time Frame: week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: days
Arm/Group | High Intensity (HI) | Low Intensity (LI)
Number analyzed (Participants) | 17 | 16
days | 62.65 (23.82) | 53.44 (33.66)

12. Other Pre Specified Outcome: Hyperpigmentation of "Normal Skin Areas" Surrounding the Target Area Exposed to Blue Light and Control Area Not Exposed to Blue Light- Evaluation by Mexameter
Description: Arbitrary units measured by mexameter. Mexameter readings ranged from 0 to 100. Higher values correspond to higher pigmentation levels.
Time Frame: week 4, 12, 16
Population: Safety Set (SAF)
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | High Intensity (HI) | Control (HI) | Low Intensity (LI) | Control (LI)
Number analyzed (Participants) | 24 | 24 | 23 | 23
arbitrary units
  4 weeks | 25.88 (6.02) | 26.58 (6.80) | 25.09 (7.86) | 23.48 (5.69)
  12 weeks | 27.71 (6.75) | 25.17 (4.65) | 24.50 (6.81) | 24.18 (5.88)
  16 weeks | 27.17 (8.61) | 26.39 (5.99) | 25.05 (6.45) | 22.95 (6.22)

13. Other Pre Specified Outcome: Adverse Events (Serious and Non-serious)
Time Frame: week 0, 1, 2, 4, 8, 12, 16
Population: Safety Set (SAF)
Measure: Number; unit: number of participants
Arm/Group | High Intensity (HI) | Low Intensity (LI)
Number analyzed (Participants) | 24 | 23
number of participants
  adverse events | 11 | 8
  serious adverse events | 0 | 0

14. Secondary Outcome: Adverse Device Events (Serious and Non-serious)
Description: Adverse device events: Adverse event related to the use of an investigational medical device wich led to any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons.
  Serious adverse device event: Adverse device effect that has resulted in a) led to death, b) led to serious deterioration in the health of the subject, that either resulted in 1) a life-threatening illness or injury, or 2) a permanent impairment of a body structure or a body function, or 3) in-patient or prolonged hospitalization, or 4) medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function, c) led to foetal distress, foetal death or a congenital abnormality or birth defect.
Time Frame: week 0, 1, 2, 4, 8, 12, 16
Population: Safety Set (SAF)
Measure: Number; unit: number of participants
Arm/Group | High Intensity (HI) | Low Intensity (LI)
Number analyzed (Participants) | 24 | 23
number of participants
  non serious | 0 | 0
  serious | 0 | 0

15. Other Pre Specified Outcome: Thermal Comfort
Description: Questionaire
Time Frame: week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | High Intensity (HI) | Low Intensity (LI)
Number analyzed (Participants) | 24 | 23
percentage of participants
  Very uncomfortable | 0.00 | 0.00
  Uncomfortable | 0.00 | 0.00
  A little uncomfortable | 4.17 | 8.70
  Just right | 25.00 | 30.43
  A little comfortable | 4.17 | 8.70
  Comfortable | 58.33 | 47.83
  Very comfortable | 8.33 | 0.00
  Missing | 0.00 | 4.35

16. Other Pre Specified Outcome: Patient Acceptance of Hyperpigmentation
Description: Questionaire
Time Frame: week 16
Population: Safety set (SAF)
Measure: Number; unit: percentage of participants
Arm/Group | High Intensity (HI) | Low Intensity (LI)
Number analyzed (Participants) | 24 | 23
percentage of participants
  Acceptable | 50.00 | 47.83
  No Hyperpigmentation | 41.67 | 47.83
  missing data | 8.33 | 4.34

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | High Intensity (HI) | Low Intensity (LI)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 11/24 | 8/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Intensity (HI) (N=24) | Low Intensity (LI) (N=23)
tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Sinobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Knee operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No